CLINICAL TRIAL: NCT01130012
Title: Feasibility of a Lifestyle Intervention in Early Risk Pregnancy in Preventing Deterioration in Glucose Tolerance?
Brief Title: Prevention of Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: South Ostrobothnia Hospital District (Unknown)
Responsible Party: Leo Niskanen PhD Prof, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KUH16032005
Record Dates: First submitted 2010-05-11; First posted 2010-05-25 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-12

CONDITIONS: Gestational Diabetes
Keywords: Gestational diabetes mellitus; Lifestyle intervention; Oral glucose tolerance test; Insulin treatment; Pregnancy outcomes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Exercise

ARMS (2):
- Lifestyle, follow-up, early care, standard care high/low risk (Other): Lifestyle: The women received counseling by a clinical nutritionist six times and by a physiotherapist six times during pregnancy.
  Interventions: Behavioral: Lifestyle: diet and exercise
- Close follow-up (Other): Follow-up: The women received information of the results of a glucose tolerance test (OGTT), reported food records three times during pregnancy, exercise history and exercise diaries monthly.
  Interventions: Behavioral: Close follow-up: reporting diaries of food and exercise

INTERVENTIONS:
Behavioral: Lifestyle: diet and exercise — Lifestyle: The women received counseling by a clinical nutritionist six times and by a physiotherapist six times during pregnancy.
  Arms: Lifestyle, follow-up, early care, standard care high/low risk
Behavioral: Close follow-up: reporting diaries of food and exercise — Follow-up: The women received information of the results of a glucose tolerance test (OGTT), reported food records three times during pregnancy, exercise history and exercise diaries monthly.
  Arms: Close follow-up

SUMMARY:
Gestational diabetes mellitus (GDM)is a major health problem

* growing prevalence of obesity
* the older age of pregnant women

A randomized controlled trial in 54 pregnant voluntary women at high risk for GDM.

* feasibility of an early intervention
* glucose tolerance at weeks 26-28

DETAILED DESCRIPTION:
1. A 75-g oral glucose tolerance test (OGTT) was performed at weeks 8-12

   1. voluntary women in early pregnancy (n=96)
   2. 54 high risk mothers were randomized

      * lifestyle intervention group (n=27)
      * close follow-up (n=27)
2. An OGTT was performed again at weeks 26-28

   * the lifestyle intervention group (n=27)
   * the close follow-up group (n=27)
   * other high-risk women of the early care group (n=42)who were not randomized
3. An OGTT was also performed at weeks 26-28 in two neighboring municipalities

   * a standard care high-risk group(n=171)who did not undergo early intervention
4. Primary outcomes

   * number of at risk participants developing GDM during pregnancy in the two arms
5. Secondary outcomes

   * the effect of intervention on fetal growth

ELIGIBILITY:
Inclusion Criteria:

* high risk for gestational diabetes
* fasting glucose 4.8-5.5 mmol/l and 2-hour glucose of OGTT <7.8 mmol/l

Exclusion Criteria:

* normal glucose tolerance at weeks 8-12
* gestational diabetes at weeks 8-12

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2005-04; Primary Completion 2006-05 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Number of at risk participants developing GDM during pregnancy

SECONDARY OUTCOMES:
The effect of intervention on fetal growth

CONTACTS AND LOCATIONS:
Overall Officials: Eeva Korpi-Hyövälti, MD, Principal Investigator — South Ostrobothnia Hospital District

REFERENCES:
- [Derived] Korpi-Hyovalti E, Heinonen S, Schwab U, Laaksonen DE, Niskanen L. Effect of intensive counselling on physical activity in pregnant women at high risk for gestational diabetes mellitus. A clinical study in primary care. Prim Care Diabetes. 2012 Dec;6(4):261-8. doi: 10.1016/j.pcd.2012.07.004. Epub 2012 Aug 13. PMID 22898328
- [Derived] Korpi-Hyovalti EA, Laaksonen DE, Schwab US, Vanhapiha TH, Vihla KR, Heinonen ST, Niskanen LK. Feasibility of a lifestyle intervention in early pregnancy to prevent deterioration of glucose tolerance. BMC Public Health. 2011 Mar 24;11:179. doi: 10.1186/1471-2458-11-179. PMID 21429234